CLINICAL TRIAL: NCT05711017
Title: The Effect of Huashibaidu Granule on Community-acquired Pneumonia in Children: a Randomized, Double-blind, Placebo-controlled Trial
Brief Title: The Effect of Huashibaidu Granule on Community-acquired Pneumonia in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Children's Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: SCMCIRB- K2022168-2
Record Dates: First submitted 2022-12-20; First posted 2023-02-02 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2022-12

CONDITIONS: Community-acquired Pneumonia
Keywords: Pediatric; community-acquired pneumonia; Huashibaidu granule
MeSH Terms: conditions — Community-Acquired Pneumonia

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Huashibaidu (Experimental): During the study, subjects diagnosed as community-acquired pneumonia in children according to "Guideline for diagnosis and treatment of community-acquired pneumonia in Children (2019 version)" will be assigned to the Huashibaidu group and the placebo group. Then they will receive 5 days treatment, prescribed by investigator according to study design. At the same time, they will finish a series of examinations, including biomarkers associated with infection, screening of pathogen, imaging examination and tNGS.
  Interventions: Drug: Huashibaidu granule
- Placebo (Placebo Comparator): During the study, subjects diagnosed as community-acquired pneumonia in children according to "Guideline for diagnosis and treatment of community-acquired pneumonia in Children (2019 version)" will be assigned to the Huashibaidu group and the placebo group. Then they will receive 5 days treatment, prescribed by investigator according to study design. At the same time, they will finish a series of examinations, including biomarkers associated with infection, screening of pathogen, imaging examination and tNGS.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Huashibaidu granule — Subjects diagnosed as community-acquired pneumonia in children at Shanghai Children's Medical Center will be consecutively screened and eligible patients will be recruited (enrolment day, day 0). The subject assigned to the Huashibaidu group will receive Huashibaidu granule two times a day for five consecutive days (day 1~5).
  Other Names: study-specified community-associated pneumonia in children drug program
  Arms: Huashibaidu
Drug: Placebo — Subjects diagnosed as community-acquired pneumonia in children at Shanghai Children's Medical Center will be consecutively screened and eligible patients will be recruited (enrolment day, day 0). The subject assigned to the placebo group will receive placebo two times a day for five consecutive days (day 1~5).
  Other Names: study-specified community-associated pneumonia in children drug program
  Arms: Placebo

SUMMARY:
The primary purpose of this study is to assess the efficacy and safety of Huashibaidu granule for the treatment of community-acquired pneumonia in children compared with placebo and to demonstrate the efficacy of Huashibaidu granule in improving clinical symptoms, removing pathogens, and shortening clinical course.

DETAILED DESCRIPTION:
Subjects diagnosed as community-acquired pneumonia in children according to "Guideline for diagnosis and treatment of community-acquired pneumonia in Children (2019 version)" at Shanghai Children's Medical Center will be consecutively screened and eligible patients will be recruited. For each enrolled patient, basic information as well as basic medical condition will be collected by investigators. The subjects will be randomly assigned to the Huashibaidu group and the placebo group.

During the study, patients will receive Huashibaidu granule or placebo two times a day for five consecutive days. Both groups of patients will receive conventional Western medical observation and symptomatic treatment, including empiric anti-infective therapy (antibiotics) and symptomatic treatment such as antipyretic, expectorant and asthmatic. Do not use other traditional Chinese medicines, proprietary Chinese medicines, and antiviral drugs. Expectorants other than Ambroxol cannot be used.

After enrollment, investigator will evaluate and score patients' clinical symptoms at day 0, 1, 2, 3, 4, 5. Detection of biomarkers associated with infection, screening of pathogen and imaging examination will be conducted at day 0. And pharyngeal swab will be collected by investigator for tNGS at day 0, 3, 5.

ELIGIBILITY:
Inclusion Criteria:

1. Han nationality.
2. Diagnosed as community-associated pneumonia in children according to "Guideline for diagnosis and treatment of community-acquired pneumonia in Children (2019 version)".
3. The first dose was given < 5 days from the onset of pneumonia (onset time is defined as the time of the first symptoms or signs of lower respiratory tract infection).
4. The guardian agrees to participate in the study and signs the informed consent form.

Exclusion Criteria:

1. The subject has severe respiratory distress, cyanosis, consciousness disorder, refusal to eat or dehydration.
2. The subject has chronic respiratory diseases, airway malformations, congenital heart disease, immune system diseases and other serious underlying diseases other than asthma.
3. The subject has moderate to severe persistent asthma or is in the acute asthma exacerbation.
4. The subject with influenza virus, pertussis, tuberculosis, fungi, and parasitic infections.
5. The subject with alanine aminotransferase (ALT) or aspartate aminotransferase (AST) 1.5 times higher than normal values in blood biochemical detection items, abnormal renal function, or troponin.
6. The subject with any other reason that investigators consider unsuitable to participate in this study.

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in clinical symptom score from baseline on day 3 | 3 days
  Investigators will compare the change of clinical symptom score from baseline on day 3 in the Huashibaidu group to the placebo group. The main symptoms assessed by the investigators are body temperature (ear temperature), daytime cough, nocturnal cough, productive sputum, thick sputum, wheezing, and shortness of breath; Secondary symptoms include dry stools, decreased appetite, poor spirit, fatigue, and diarrhoea. Each symptom is assigned a score of 0, 1, 2, and 3 by investigators according to the symptoms from mild to severe.

SECONDARY OUTCOMES:
Anti-infective efficacy of Huashibaidu granule | 5 days
  Investigators will collect throat swabs from subjects for targeted next-generation sequencing (tNGS) detection to compare the change of pathogen sequence numbers from baseline on day 3 and day 5 in the Huashibaidu group to the placebo group.There are 95 target pathogens, including 31 DNA viruses, 38 RNA viruses, 10 gram-positive bacteria, 12 gram-negative bacteria, 1 mycoplasma and 3 chlamydia. For example, human adenovirus (23 species), human herpesvirus (5 species), enterovirus (6 species), coxsackievirus (5 species), human coronavirus (4 species), human respiratory syncytial virus (2 species) and so on.
time to symptom resolution | 5 days
  Subjects will be scored daily for pneumonia symptom. And investigators will compare the time to pneumonia symptom resolution in the Huashibaidu group to the placebo group.
total effective rate | 5 days
  Efficacy index (%) = {(symptom score before treatment - symptom score after treatment) / symptom score before treatment} * 100%. Significant efficiency: efficacy index greater than equal to or equal to 70%. Efficiency: efficacy index greater than or equal to 30% but less than 70%. Total effective rate = significant efficiency + effective rate.
change on the number of different pathogens sequences | 5 days
  Investigators will record the change on the number of different pathogens sequences in the Huashibaidu group and the placebo group.
changes in cytokines | 5 days
  Investigators will record the change in cytokines in the Huashibaidu group and the placebo group, which contain IL-1β, IL-4, IL-5, IL-6, IL-8, IL-17a, IL-12, IL-13, TGF-β1, IFN-α, IFN-β, IFN-γ, TNF-α, TNF-β and ISG-15.
Duration of hospitalization | 5 days
  Investigators will compare the duration of hospitalization in the Huashibaidu group to the placebo group.
Rate of transition to severe pneumonia | 5 days
  Rate of transition to severe pneumonia = number of subjects who have turned severe pneumonia / total number of subjects in the Huashibaidu group or placebo group.
Rate of transition to ICU | 5 days
  Rate of transition to ICU = number of subjects who have been transferred from the general ward to the ICU / total number of subjects in the Huashibaidu group or placebo group.

CONTACTS AND LOCATIONS:
Overall Officials: Yong Yin, PhD, Principal Investigator — Shanghai Children's Medical Center

IPD SHARING:
Plan to Share IPD: No